CLINICAL TRIAL: NCT02261649
Title: The Impact of Cerebellar Mass Resection on Pain Processing
Brief Title: Impact of Cerebellar Mass Resection on Pain Processing
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric Moulton, PhD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 14-104; 1R21CA185870-01 (NIH)
Record Dates: First submitted 2014-10-02; First posted 2014-10-10 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Cerebellar Neoplasm
Keywords: Cerebellar tumor; Non-malignant low-grade cerebellar astrocytomas
MeSH Terms: conditions — Cerebellar Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cerebellar Tumor Surgically Removed: Quantitative Sensory Testing and Neuroimaging
  * Medoc Advanced Medical Systems PATHWAY Model ATS (Contact thermal stimulator)
  * Cold water bath
  * MRI scanner
  * Questionnaires
  Interventions: Device: Medoc Advanced Medical Systems PATHWAY Model ATS; Procedure: Cold water bath; Device: MRI scanner; Other: Questionnaires
- Healthy Volunteer: Quantitative Sensory Testing and Neuroimaging
  * Medoc Advanced Medical Systems PATHWAY Model ATS (Contact thermal stimulator)
  * Cold water bath
  * MRI scanner
  * Questionnaires
  Interventions: Device: Medoc Advanced Medical Systems PATHWAY Model ATS; Procedure: Cold water bath; Device: MRI scanner; Other: Questionnaires

INTERVENTIONS:
Device: Medoc Advanced Medical Systems PATHWAY Model ATS — 30 minutes of sensory testing using a contact thermal stimulator will measure thresholds for heat and cool detection, and threshold for hot and cold pain.
Procedure: Cold water bath — The next 15 minutes of sensory testing will measure tolerance to having right or left hand in a tub of cold water. The participant will place their hand in cold water and leave it there for as long they can, even if it is uncomfortable. The participant can take their arm out if it gets too uncomfortable to leave it in.
Device: MRI scanner — An MRI will be used to collect anatomical and functional images from patients and subjects. These data will be collected within a 1 hour block.
Other: Questionnaires — The surveys include questions about emotions, thoughts, and feelings. These surveys will be given before sensory testing and before the MRI scan. The parent or guardian will help to complete two surveys, and will complete one survey on his or her own. Questions can be skipped, and may be stopped at any time.

SUMMARY:
The purpose of the study is to evaluate how cerebellar resection surgery may affect pain sensation and the way the brain "reads" pain signals. By measuring brain activity in children and adolescents following surgery, the investigators hope to gain valuable information about pain processing in the brain.

DETAILED DESCRIPTION:
This study is designed to test whether cerebellar resection surgery affects pain pathways in the brain. To participate a participant must (A) have had a cerebellar mass surgically removed, or (B) are a healthy volunteer with no history of pain disorders or mental illness. The study will involve sensory testing and brain imaging using magnetic resonance imaging (MRI) Sensory testing will be performed using a tub of cold water, as well as a contact thermode capable of delivering hot and cold temperatures. MRI brain scanning uses magnetic fields and radio waves to give pictures of the brain without using radiation.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age 4-18 years old at the time of surgery
* Resection limited to the cerebellum
* Within 20 years of surgery
* Good physical health excluding symptoms directly related to cerebellar resection
* No cerebellar-mass directed treatment other than surgical resection

Inclusion Criteria for all subjects:

* Age 6-38 years old at the time of participation
* No paralysis/hemiparesis
* No motor deficits that would interfere with performance or required tasks (button press withdraw hand from water bath)
* English speaking sufficient to comprehend and provide assent with parental assistance or consent if over the age of 18
* Ability to complete MRI without sedation

Exclusion Criteria:

* Claustrophobia
* Significant medical (e.g. asthma, renal, cardiac, gastrointestinal or immunological) or brain- related disorders (e.g. seizures, autism, psychiatric conditions such as severe depression, psychosis)
* Metallic or magnetic implants that pose a risk to the participant or to the data quality
* Weight > 285 pounds (weight limit of the fMRI table)
* History of drug abuse or positive drug screen
* Positive pregnancy screen
* Use of antidepressants or anticonvulsants, excepting patient usage after resection
* Significant alcohol history (ingestion of 5 or more glasses (> 40 oz) of alcohol per week)
* Tattoos containing metallic ink on the neck, shoulders, upper arm and head (which could heat up in the scanner, and potentially cause blistering or burning)
* Cardiac pacemakers
* Aneurysm clips and other vascular stents, filters, clips or other devices
* Prosthetic heart valves
* Other prostheses
* Neuro-stimulator devices
* Implanted infusion pumps
* Cochlear (ear) implants
* Ocular (eye) implants or known metal fragments in eyes
* Exposure to shrapnel or metal filings (sheet metal workers, welders, and others)
* Participants that require anesthesia to complete an MRI scan
* Receipt of a medication via transdermal patch

Ages: 6 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with cerebellar resection and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Increase in blood oxygen level dependent signal response | Baseline, Day 1
  Functional magnetic resonance imaging scans will be collected to measure blood oxygen level dependent (BOLD) responses, an indirect measure measure of neural activity. The Unit of Measure is % BOLD signal change across spatiotemporal domains within the brain.

SECONDARY OUTCOMES:
Fear of Pain Questionnaire-Child scores | Baseline, Day 1
  Assesses fear of pain
Multidimensional Anxiety Scale for Children scores | Baseline, Day 1
  Assesses anxiety
Behavior Rating Inventory of Executive Function scores | Baseline, Day 1
  Assesses executive function
Fear of Pain Questionnaire III-Adult scores | Baseline, Day 1
  Assesses fear of pain
Multidimensional Anxiety Questionnaire-Adult scores | Baseline, Day 1
  Assesses anxiety
Behavior Rating Inventory of Executive Function-Adult version scores | Baseline, Day 1
  Assesses executive function

CONTACTS AND LOCATIONS:
Overall Officials: Eric Moulton, Ph.D, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Waltham, Massachusetts, United States